CLINICAL TRIAL: NCT00841113
Title: Phase III Study of the Comparison of Abarelix Versus Goserelin Plus Bicalutamide in Patients With Advanced or Metastatic Prostate Cancer. A One Year Randomised, Open Label, Multi-Centre Phase III Trial.
Brief Title: Abarelix Versus Goserelin Plus Bicalutamide in Patients With Advanced or Metastatic Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Speciality European Pharma Limited (Industry)
Responsible Party: Speciality European Pharma Limited, SEP
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABACAS1
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2009-02-11 (Estimated); Status verified 2009-02

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Advanced; Metastatic
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — abarelix; Goserelin; bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Abarelix (Experimental): Investigative drug
  Interventions: Drug: Abarelix
- 2 Goserelin plus bicalutamide (Active Comparator): Standard therapy
  Interventions: Drug: Goserelin plus Bicalutamide

INTERVENTIONS:
Drug: Abarelix — 100 mg by Intramuscular injection on days; 1, 15 and 29 and monthly thereafter
  Other Names: Plenaxis
  Arms: 1 Abarelix
Drug: Goserelin plus Bicalutamide — Goserelin - 3.6 mg by monthly subcutaneous injection Biaclutamide 50 mg orally daily for first three months
  Arms: 2 Goserelin plus bicalutamide

SUMMARY:
To compare the safety of efficacy of abarelix versus goserelin plus bicalutamide in patients with advanced or metastatic prostate cancer.

DETAILED DESCRIPTION:
Inclusion Criteria

* Males over 18 with documented advanced or metastatic prostate cancer

Outcome measures

* Comparative castration rates one week after starting therapy
* Degree of testosterone surge in the first month of treatment.
* Maintenance of medical castration during one year of therapy.
* Comparison of the treatments on QTc prolongation

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven prostate cancer and not previously treated with hormones
* Evidance of advanced disease or metastases
* Life expentancy of at least 3 months
* Normal serum testosterone levels
* Written informed consent

Exclusion Criteria:

* Previous endocrine or cytoxic theapy for prostate cancer
* Known tumour complication of prostate cancer which owuld require immediate treatment
* Another malignancy other than basal cell cancer
* History of significant drug hypersensitivity to either LHRH agonists or GnRH antagonists.
* Congenital or acquired coagulation disorders contraindicating intramuscular injections
* Pagets disease of the bone
* QTcB > 450 msec at Day - 14

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 1999-01; Primary Completion 2001-02 (Actual); Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
Early castration rates | One week

SECONDARY OUTCOMES:
Maintenance of medical castration | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Frans M J Debruyne, MD, Principal Investigator — University Hospital Nijmegen